CLINICAL TRIAL: NCT05250947
Title: A Phase I Study Evaluating the Safety and Feasibility of Platelet-rich Plasma for the Treatment of Facetogenic Low Back Pain
Brief Title: Study Evaluating the Safety and Feasibility of Platelet-rich Plasma to Treat Facetogenic Low Back Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Projected cost to continue was not supported by the study budget and additional funds could not be obtained so the decision to close the study was made.
Sponsor: Matthew Pingree (Other)
Responsible Party: Sponsor-Investigator, Matthew Pingree, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-011475
Record Dates: First submitted 2022-01-04; First posted 2022-02-22 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Spondylosis
Keywords: arthritis; facet joint; lumbar spondylosis; back pain
MeSH Terms: conditions — Spondylosis; Arthritis; Back Pain

STUDY DESIGN:
Intervention Model Description: This is a pilot safety study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- PRP Injection Arm (Experimental): The FDA cleared Angel® Concentrated Platelet Rich Plasma System and Angel® cPRP Processing Set will be used to process the PRP. The targeted final PRP volume of 6 ml will be injected in up to 4 facet joints (2 levels) at 1.5 ml per joint.
  Interventions: Device: Angel® Concentrated Platelet Rich Plasma System; Drug: Platelet Rich Plasma

INTERVENTIONS:
Device: Angel® Concentrated Platelet Rich Plasma System — Angel® Concentrated Platelet Rich Plasma System and Angel® cPRP Processing Set will be used to process the PRP.
Drug: Platelet Rich Plasma — 6 ml will be injected in up to 4 facet joints (2 levels) at 1.5 ml per joint

SUMMARY:
This study is being done to assess the safety of using the Angel Concentrated Platelet Rich Plasma System to process Platelet Rich Plasma (PRP) to treat arthritis of the low back (lumbar spondylosis).

DETAILED DESCRIPTION:
This study is a pilot of the safety of using the FDA cleared Angel® Concentrated Platelet Rich Plasma System and Angel® cPRP Processing Set to process PRP to treat arthritis of the low back (lumbar spondylosis). Subjects will be screened at outpatient clinic visit appointments and interested qualified subjects will be consented and offered participation in this trial. Once consent has been obtained baseline values will be established and subjects will begin treatment and follow-up for the next 12 months. A final visit for evaluation and collection of lab samples will be conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiographic (MRI, CT or lumbar x-ray) evidence of symptomatic facet arthropathy involving the bilateral bottom two facets (e.g., L4-5 or L5-6 and L5-S1 or L6-S1).
* Positive response, defined according to current clinical standards for the diagnosis of facet-mediated low back pain as greater than or equal to 75% pain improvement (as reported by patient) to diagnostic medial branch nerve blocks, one block with lidocaine and the other with bupivacaine.
* Low back pain VAS score of greater than or equal to 5 at the clinical visit just prior to the first medial branch nerve block.

Exclusion Criteria:

* Prior facet related procedure (intraarticular corticosteroid injection, radiofrequency ablation (RFA)) in last 6 months or prior fusion in the bottom two facets.
* Current opioid use of greater than 50mg oral morphine milligram equivalents per day.
* No advanced imaging (MRI, CT or lumbar x-ray) of the lumbar spine within the last 6 months.
* BMI > 34.99 (WHO class I obesity).
* Active systemic or local infection as evidenced by fever >100.4 degrees Fahrenheit, or any other clinical signs or symptoms of infection within 24 hours of the procedure.
* On anticoagulation drug and has been on hold for less than 7 days prior to the investigational procedure.
* Imaging evidence of high likelihood of failure for intra-articular injection in the opinion of the PI or delegate review of MRI, CT or lumbar x-ray imaging.
* History of chronic thrombocytopenia (or pre-operative platelet count less than 195,000 per μl).
* Undergoing chemotherapy at time of injection.
* Pregnant or breastfeeding.
* Use of illicit drugs within 30 days prior to study entry.
* NSAID use during the pre-procedural period (one week before Treatment Day 0).
* Preoperative hematocrit less than 36%.
* History of hemodynamic instability or inability to maintain stable oncotic pressure.
* History of prolonged clotting times.
* Prior history of lumbar procedure.
* Redness, swelling, rash or other concerning lesions at the injection site just prior to the procedure.
* Prior history of allergy to lidocaine or other local anesthetic agent.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Number of adverse device effects | Day 0 (Day of procedure)
  Adverse device effects related to the processing of the platelet rich plasma product (such as hardware failures/malfunctions, software errors, disposable set equipment malfunctions, processing errors, automatic self-test/calibration errors, variations in hematocrit level in final product, variations in total volume of PRP concentrate produced, etc.)
Number of suspected acute adverse reactions to the treatment | Day 0 to Day 14
  Suspected adverse reactions to the treatment based on evaluations including follow-up physical examinations, labs and assessment of clinical signs and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Pingree, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No